CLINICAL TRIAL: NCT02834312
Title: A Multicentre Dose-Finding, Randomised, Double-Blind, Placebo-Controlled Study to Select the Daily Oral Dose of Estetrol (E4) for the Treatment of Vasomotor Symptoms in Post-Menopausal Women
Brief Title: E4Relief (Response to Estetrol in Life Improvement for MEnopausal-associated Hot Flushes)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Donesta Bioscience (Industry)
Collaborators: SynteractHCR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIT-Do0001-C201; 2015-004018-44 (EudraCT Number)
Record Dates: First submitted 2016-07-07; First posted 2016-07-15 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Hot Flushes
Keywords: Estetrol; Vasomotor symptoms; Menopause
MeSH Terms: conditions — Hot Flashes | interventions — Estetrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 2.5 mg estetrol (Experimental)
  Interventions: Drug: Estetrol
- 5 mg estetrol (Experimental)
  Interventions: Drug: Estetrol
- 10 mg estetrol (Experimental)
  Interventions: Drug: Estetrol
- 15 mg estetrol (Experimental)
  Interventions: Drug: Estetrol
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estetrol — All treatments (E4 [2.5 mg, 5 mg, 10 mg, 15 mg] capsule) will be administered once daily (QD) per os for at least 12 consecutive weeks until the last biological assessments (Day 90 maximum) have been performed.
  Other Names: E4
  Arms: 10 mg estetrol; 15 mg estetrol; 2.5 mg estetrol; 5 mg estetrol
Drug: Placebo — 1 capsule will be administered QD per os for at least 12 consecutive weeks until the last biological assessments (Day 90 maximum) have been performed.
  Arms: placebo

SUMMARY:
This dose-finding study is being conducted to select the daily oral dose of estetrol (E4) for the treatment of vasomotor symptoms (VMS) in post-menopausal women.

DETAILED DESCRIPTION:
Oestrogen therapy is the most consistently effective treatment used in the US and Europe for menopausal VMS. Following the safety issues reported in the primary Women's Health Initiative publications and with continued subject requests for treatment, a challenge to clinicians has been to identify the lowest effective dose of oestrogen for alleviating menopausal symptoms. In addition, it is a challenge to develop a safer oestrogen than those currently used.

For this purpose, the minimum effective dose (MED) of E4 has to be defined for the treatment of menopausal symptoms. The present study is intended to evaluate changes in frequency and in severity of moderate to severe VMS in order to define the MED.

Subjects will be randomly allocated to either treatment group (2.5 mg E4, 5 mg E4, 10 mg E4, 15 mg E4, or placebo) in a 1:1:1:1:1 ratio. All treatments (E4 or Placebo) will be administered once daily (QD) per os for at least 12 consecutive weeks until the last biological assessments (Day 90 maximum) have been performed.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting at least 7 moderate to severe hot flushes/day or at least 50 moderate to severe hot flushes/week in the week preceding randomization.
* Body Mass Index (BMI) between 18.0 and 35.0 kg/m², inclusive.
* Post-menopausal status.
* Intact uterus.
* Negative pregnancy test.
* Good physical and mental health.
* Subject has provided signed and dated written informed consent before admission to the study.
* Subject is able to understand and comply with the protocol requirements, instructions, and protocol-stated restrictions.

Exclusion Criteria:

* Uterine disease or any medical conditions associated with an increase in endometrial thickness.
* Any history of malignancy with the exception of basal cell (excluded if within the prior 2 years) or squamous cell (excluded if within the prior one year) carcinoma of the skin. Any clinically significant findings at the breast examination and/or on mammography suspicious of breast malignancy that would require additional clinical testing to rule out breast cancer.
* Abnormal cervical Pap smear.
* Systolic blood pressure (BP) outside the range 90 to 140 mmHg, diastolic BP outside the range 60 to 90 mmHg, and/or heart rate outside the range 40 to 100 bpm.
* Any clinically significant abnormality identified on the screening 12-lead ECG.
* History of venous or arterial thromboembolic disease, history of known coagulopathy or abnormal coagulation factors.
* Diabetes mellitus with poor glycaemic control.
* Dyslipoproteinaemia at screening.
* Smoking >10 cigarettes/day.
* Presence or history of gallbladder disease, unless cholecystectomy has been performed.
* Systemic lupus erythematosus.
* Multiple sclerosis.
* Acute or chronic liver disease.
* Acute or chronic renal impairment.
* Uncontrolled thyroid disorders.
* Use of oestrogen or progestin containing drug(s).
* Use of non-hormonal treatments to reduce hot flushes.
* History or presence of allergy or intolerance to any component of the investigational product.
* History of alcohol or substance abuse or dependence in the 12 months before screening as determined by the Investigator.
* Sponsor, CRO or Investigator's site personnel or their relatives directly affiliated with this study.
* Subjects with known or suspected history of a clinically significant systemic diseases, unstable medical disorders, life-threatening disease or current malignancies that would pose a risk to the subject in the opinion of the Investigator.
* Participation in another investigational drug clinical study within 1 month (30 days) or have received an investigational drug within the last 3 months (90 days) prior to study entry.
* Is judged by the Investigator to be unsuitable for any reason.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Change in weekly frequency of moderate to severe VMS from baseline to week 4. | From baseline to week 4
Change in weekly frequency of moderate to severe VMS from baseline to week 12. | From baseline to week 12
Change in severity of moderate to severe VMS from baseline to week 4. | From baseline to week 4
  The Severity Scoring System of VMS will be documented by the subjects by using the following scores:
  None (0) = No VMS symptoms; Mild (1) = Sensation of heat without sweating; Moderate (2) = Sensation of heat with sweating. Able to continue activity; Severe (3) = Sensation of heat with sweating. Causes cessation of activity.
Change in severity of moderate to severe VMS from baseline to week 12. | From baseline to week 12
  The Severity Scoring System of VMS will be documented by the subjects by using the following scores:
  None (0) = No VMS symptoms; Mild (1) = Sensation of heat without sweating; Moderate (2) = Sensation of heat with sweating. Able to continue activity; Severe (3) = Sensation of heat with sweating. Causes cessation of activity.

SECONDARY OUTCOMES:
Change from baseline to week 12 in genitourinary symptoms (GSM) of menopause | From baseline to week 12
  The following GSM symptoms will be evaluated:
  * Vaginal dryness (none, mild, moderate or severe)
  * Vaginal and/or vulvar irritation/itching (none, mild, moderate or severe)
  * Dysuria (none, mild, moderate or severe)
  * Vaginal pain associated with sexual activity (none, mild, moderate or severe)
  * Vaginal bleeding associated with sexual activity (presence vs. absence).
Change in the Menopause Rating Scale (MRS) from baseline to week 5. | From baseline to week 5
Change in the Menopause Rating Scale (MRS) from baseline to week 12. | From baseline to week 12
Change from baseline to week 12 in Vaginal pH. | From baseline to week 12
Change from baseline to week 12 in Vaginal Maturation Index (MI) (parabasal and superficial cells) | From baseline to week 12
Serum concentration of triglycerides. | From baseline to week 12
Serum concentration of low density lipoprotein (LDL)-cholesterol. | Baseline and Week 12
Serum concentration of high density lipoprotein (HLD)-cholesterol. | Baseline and Week 12
Serum concentration of total cholesterol. | Baseline and Week 12
Fasting glycemia. | Baseline and Week 12
Serum concentration of glycated hemoglobin. | Baseline and Week 12
Homeostasis model assessment-estimated insulin resistance [HOMA-IR] | Baseline and Week 12
Serum concentration of prothrombin fragment 1 + 2. | Baseline and Week 12
Activated protein C sensitivity ratio (APCsr) (Endogenous Thrombin Potential [ETP]-Based). | Baseline and Week 12
Serum concentration of D-dimers. | Baseline and Week 12
Serum concentration of sex-hormone binding globulin (SHBG). | Baseline and Week 12
Serum concentration of antithrombin. | Baseline and Week 12
Serum concentration of protein-C. | Baseline and Week 12
Serum concentration of free protein-S. | Baseline and Week 12
Serum concentration of factor VIII. | Baseline and Week 12
Serum concentration of free tissue factor pathway inhibitor [TFPI]. | Baseline and Week 12
Serum concentration of osteocalcin. | Baseline and Week 12
Serum concentration of C-terminal telopeptide [CTX-1] | Baseline and Week 12
Percentage of subjects who had a change in endometrial thickness at each study visit. | From baseline to week 16
Percentage of subjects with adverse events as a measure of safety and tolerability. | Up to week 16
Maximum concentration (Cmax) of E4 in plasma. | Up to 90 days
Time to Cmax (Tmax) of E4 in plasma. | Up to 90 days
Terminal half-life (T1/2) of E4 in plasma. | Up to 90 days
Area under the plasma concentration-time curve from baseline to the last quantifiable concentration following dosing (AUCtau) of E4. | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Donesta Bioscience, Study Director — Donesta Bioscience BV
Locations (1):
- Donesta Bioscience BV, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaspard U, Taziaux M, Jost M, Coelingh Bennink HJT, Utian WH, Lobo RA, Foidart JM. A multicenter, randomized, placebo-controlled study to select the minimum effective dose of estetrol in postmenopausal participants (E4Relief): part 2-vaginal cytology, genitourinary syndrome of menopause, and health-related quality of life. Menopause. 2023 May 1;30(5):480-489. doi: 10.1097/GME.0000000000002167. Epub 2023 Feb 20. PMID 36809193
- See also: Trial results were released to public view on the EudraCT (EudraCT Number: 2015-004018-44). — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-004018-44/results